CLINICAL TRIAL: NCT03749811
Title: Comparison of Remifentanil Consumption in Pupillometry-guided Versus Conventional Administration in Pediatric Surgery: a Prospective, Randomized Controlled Trial
Brief Title: Pupillometry-guided Remifentanil Infusion Versus Conventional Administration in Children
Acronym: PURFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, princial investigator, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1811-036-984
Record Dates: First submitted 2018-11-18; First posted 2018-11-21 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Opioid Use
Keywords: Pupil dilatory reflex; Remifentanil; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Interventional group: remifentanil infusion under pupillometry monitoring. Control group: remifentanil infusion without pupillometry monitoring (remifentanil dose is determined by conventional method, i. e., hemodynamic change probably related to noxious stimuli)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant does not know in which of the groups he/she is allocated. Only a care provider (an attending anesthesiologist who is responsible for the patient's anesthesia) knows the group which the patient belongs to.
  Investigator and outcomes assessor does not know in which of the groups the patient is allocated, since the group name will be just recorded as "A" or "B" until data analysis of the last participant is done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pupillometry group (Experimental): A group of participants who receive remifentanil infusion under pupillometry monitoring.
  Interventions: Device: Pupillometry
- Conventional group (No Intervention): A group of participants who receive remifentanil infusion without pupillometry monitoring; their analgesic dose is mainly determined via hemodyamic change.

INTERVENTIONS:
Device: Pupillometry — After induction of anesthesia and determination of the loss of consciousness of the participant, baseline diameter of pupil is measured by electronic pupillometry device. During anesthesia, participant's pupil diameter is repeatedly measured with 5-minute interval. Pupil dilation of 30% or more compared to baseline is indicative of insufficient analgesia.
  Arms: Pupillometry group

SUMMARY:
Our study aims to compare the total intravenous dose of remifentanil per anesthesia hour and body weight in two groups of pediatric surgical patients - an interventional group with remifentanil infusion under pupillometry monitoring, and control group without pupillometry - to figure out whether pupillometry monitoring may reduce remifentanil consumption during anesthesia while providing sufficient analgesia for surgical noxious stimuli.

DETAILED DESCRIPTION:
comparison of total used opioid

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients who are at 3 to 6 years of age, scheduled to undergo elective surgery with estimated time of operation 2 hours or longer, under general anesthesia
* American Society of Anesthesiologists physical status classification (ASA class) I - II
* Patient and his/her parents are willing to participate after explanation of the purpose, materials, methods, possible risks and benefits of the research

Exclusion Criteria:

* History of hypersensitivity/allergic reaction to the drugs which are used in general anesthesia
* Preoperative use of analgesics, antipsychotics and/or antiepileptics
* Mental retardation
* Medications related to hindrance of autonomic nerve system activity, e. g., beta blockers
* Underlying ophthalmic diseases

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2020-11-18 (Estimated); Study Completion 2021-11-18 (Estimated)

PRIMARY OUTCOMES:
remifentanil total dose in microgram | from beginning of anesthesia to the end of the anesthesia
  Remifentanil total dose divided by anesthesia time (minute) and patient weight (kg).
FLACC score | Arrival at the post-anesthesia care unit
  FLACC score (a pain evaluation method for children who cannot express their severity of pain verbally) right after post-anesthesia care unit arrival.
Adjusted analgesic dose after anesthesia | 24 hours after the end of anesthesia
  Total dose of analgesics (NSAIDs and opioids) delivered to the patient since the end of the anesthesia, until 24 hours after the end of anesthesia

SECONDARY OUTCOMES:
Emergence time | Intraoperative
  Time between the end of the surgery and extubation
Incidence of rescue therapy | Intraoperative
  Incidence of vasopressor/inotropics/anticholinergics/fluid/vasodilators administered, due to moderate to severe hemodynamic change

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D., Ph.D., Principal Investigator — Dept. of Anesthesiology and Pain Medicine, Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wildemeersch D, Peeters N, Saldien V, Vercauteren M, Hans G. Pain assessment by pupil dilation reflex in response to noxious stimulation in anaesthetized adults. Acta Anaesthesiol Scand. 2018 Sep;62(8):1050-1056. doi: 10.1111/aas.13129. Epub 2018 Apr 19. PMID 29671874
- [Result] Sabourdin N, Barrois J, Louvet N, Rigouzzo A, Guye ML, Dadure C, Constant I. Pupillometry-guided Intraoperative Remifentanil Administration versus Standard Practice Influences Opioid Use: A Randomized Study. Anesthesiology. 2017 Aug;127(2):284-292. doi: 10.1097/ALN.0000000000001705. PMID 28719527